CLINICAL TRIAL: NCT00313027
Title: Cervical Nodal Metastasis in Squamous Cell Carcinoma of the Head and Neck - Novel MRI, FDG-PET, and Histopathologic Correlation
Brief Title: Cervical Nodal Mets in Squamous Cell Carcinoma of H&N - MRI, FDG-PET, & Histopathologic Correlation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ENT0011; 78639; ENT0011; NCT00313027
Record Dates: First submitted 2006-03-27; First posted 2006-04-11 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Head and Neck Cancer; Carcinoma, Squamous Cell; Head and Neck Cancers
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Radiation: PET scan

SUMMARY:
The purpose of this study is to determine the value of novel non-invasive medical imaging methods for detecting the spread of head and neck squamous cell carcinoma to the lymph nodes in the neck by comparing their results to findings at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:- Adult patients with newly diagnosed (biopsy-proven), untreated squamous cell carcinoma (SCC) of the head and neck who will undergo neck dissection as part of primary surgical therapy. Exclusion Criteria:- A prior adverse reaction to the contrast/tracer agents being used in the imaging methods being studied.

- Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-11; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the performance of novel imaging methods for detecting cervical nodal metastasis. | pre and post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Billy W. Loo Jr. M.D. Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States